CLINICAL TRIAL: NCT02109003
Title: Efficiency of PressureEasy in Controlling Tracheal Cuff Pressure in Intubated Critically Ill Patients
Brief Title: Efficiency of a Mechanical Device in Controlling Tracheal Cuff Pressure in Intubated Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Antonio Artigas Raventós, Director of Critical Care Unit, Corporacion Parc Tauli
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EPREI
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Cuff Overinflation; Cuff Underinflation
Keywords: tracheal cuff; cuff overinflation; cuff underinflation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous control of Pcuff followed by manual control (Experimental): Patients receive continuous control of cuff pressure with Pressure easy® device for 24h, followed by discontinuous control (every 4 hours) with a manual manometer for 24 h.
  Interventions: Device: Pressure easy® device
- Manual control of Pcuff followed by continuous control. (Active Comparator): Patients receive the reverse sequence (manual control followed by continuous control of Pcuff)
  Interventions: Device: Manual control of Pcuff followed by continuous control.

INTERVENTIONS:
Device: Pressure easy® device — Continuous control of tracheal cuff pressure using a mechanical device for 24h followed by manual control of cuff pressure using a manometer.
  Other Names: Pressure easy® device (Smiths medical cuff pressure controller)
  Arms: Continuous control of Pcuff followed by manual control
Device: Manual control of Pcuff followed by continuous control. — Control 24h with manual control using a manometer followed by 24h of continuous control using a mechanical device.
  Arms: Manual control of Pcuff followed by continuous control.

SUMMARY:
Despite intermittent control of tracheal cuff pressure using a manual manometer, cuff underinflation and overinflation frequently occur in critically ill patients, resulting in increased risk for microaspiration and tracheal ischemic lesions.

DETAILED DESCRIPTION:
The aim of this study is to determine the efficiency of Pressure easy® device (Smiths medical cuff pressure controller) in continuous control of tracheal cuff pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients intubated in the ICU with a polyvinyl chloride (PVC) cuffed tracheal tube.
* Predicted duration of mechanical ventilation > or = 48h.
* Age > or = 18 years.
* Signed informed consent.

Exclusion Criteria:

* Anticipated duration of mechanical ventilation<48h after randomization.
* Tracheostomized patients.
* Patients with contraindication for semirecumbent position.
* Patients participating to another trial that might influence this study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of recording time spent with cuff overinflation or underinflation | 48 hours
  Continuous recording of cuff pressure will be performed during two 24-h periods (with or without Pressure easy® device)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Rodriguez, MD, Principal Investigator — Critical Care Unit. Hospital de Sabadell, Corporación Sanitaria y Universitaria Parc Taulí
Locations (1):
- Area de Críticos, Hospital de Sabadell, Corporación Sanitaria y Universitaria Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Nseir S, Rodriguez A, Saludes P, De Jonckheere J, Valles J, Artigas A, Martin-Loeches I. Efficiency of a mechanical device in controlling tracheal cuff pressure in intubated critically ill patients: a randomized controlled study. Ann Intensive Care. 2015 Dec;5(1):54. doi: 10.1186/s13613-015-0054-z. Epub 2015 Jun 2. PMID 26059205